CLINICAL TRIAL: NCT00842842
Title: A Prospective, Controlled, Randomized, Patient and Evaluator Blinded Study to Evaluate Pain and Recovery in Patients Undergoing Laparoscopic Umbilical Hernia Repair by Fixing the Mesh With Tisseel Versus Tackers
Brief Title: Mesh Fixation With Intraperitoneal Tisseel
Acronym: MEFIXIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Jens Ravn Eriksen, MD PhD, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-B-2008-147
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Postoperative Pain; Ventral Hernia
Keywords: surgical fixation devices; postoperative pain; ventral hernia; fibrin tissue adhesive; laparoscopy; quality of life; fatigue
MeSH Terms: conditions — Pain, Postoperative; Hernia, Ventral; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: tacks (Active Comparator): mesh fixation with tacks
  Interventions: Procedure: tack fixation of mesh
- 2: glue (Experimental): mesh fixation with glue
  Interventions: Procedure: glue fixation of mesh

INTERVENTIONS:
Procedure: tack fixation of mesh — tack fixation of mesh
  Arms: 1: tacks
Procedure: glue fixation of mesh — glue fixation of mesh
  Arms: 2: glue

SUMMARY:
The purpose of this study is to determine whether mesh fixation in laparoscopic umbilical hernia repair with fibrin glue is superior to tacks in terms of postoperative pain and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-85 years and Danish speaking
* Umbilical hernia Ø 1.5 - 5 cm at preoperative clinical examination
* ASA group I-III

Exclusion Criteria:

* Former laparoscopic umbilical herniotomy
* Incarceration
* Drug/alcohol abuse/ongoing use of strong analgesic
* Bad compliance
* Liver disease Child-Pugh stage B/C
* Immunodeficiency (ex. steroid use)
* Pregnancy
* Other hernias recognized perop. and operated on at the same operation
* Lack of consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Postoperative pain VAS 0-100 mm | 1 year

SECONDARY OUTCOMES:
QoL, SF-36, recurrence (safety) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rosenberg, Professor, D.Sc, Study Chair — Herlev University Hospital, Dept. Surg. Gastroenterology
Locations (4):
- Denmark (4):
  - Bispebjerg University Hospital, Dept. Surgical Gastroenterology, Copenhagen
  - Gentofte University Hospital, Dept. Surg. Gastroenterology, Gentofte, Copenhagen
  - Herlev University Hospital, Dept. Surgical Gastroenterology, Herlev
  - Køge University Hospital, Dept. Surg. Gastroenterology, Koege

REFERENCES:
- [Background] Eriksen JR, Poornoroozy P, Jorgensen LN, Jacobsen B, Friis-Andersen HU, Rosenberg J. Pain, quality of life and recovery after laparoscopic ventral hernia repair. Hernia. 2009 Feb;13(1):13-21. doi: 10.1007/s10029-008-0414-9. Epub 2008 Aug 1. PMID 18670733
- [Background] Eriksen JR, Bech JI, Linnemann D, Rosenberg J. Laparoscopic intraperitoneal mesh fixation with fibrin sealant (Tisseel) vs. titanium tacks: a randomised controlled experimental study in pigs. Hernia. 2008 Oct;12(5):483-91. doi: 10.1007/s10029-008-0375-z. Epub 2008 May 16. PMID 18483783
- [Background] Eriksen JR, Gogenur I, Rosenberg J. Choice of mesh for laparoscopic ventral hernia repair. Hernia. 2007 Dec;11(6):481-92. doi: 10.1007/s10029-007-0282-8. Epub 2007 Sep 11. PMID 17846703
- [Derived] Eriksen JR, Bisgaard T, Assaadzadeh S, Jorgensen LN, Rosenberg J. Randomized clinical trial of fibrin sealant versus titanium tacks for mesh fixation in laparoscopic umbilical hernia repair. Br J Surg. 2011 Nov;98(11):1537-45. doi: 10.1002/bjs.7646. Epub 2011 Aug 24. PMID 21964681